CLINICAL TRIAL: NCT07110675
Title: Identification of Central Sensitisation in Patients With Haemophilia and Degenerative Arthropathy of the Lower Limbs. A Cross-sectional Cohort Study
Brief Title: Central Sensitisation in Patients With Haemophilia and Degenerative Arthropathy
Status: Recruiting | Type: Observational
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Principal Investigator, Rubén Cuesta-Barriuso, Principal Investigator, Investigación en Hemofilia y Fisioterapia
Other Study IDs: He-Sens
Record Dates: First submitted 2025-07-25; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Hemophilia
Keywords: Hemophilia; Joint pain; Central sensitization; Disability; Kinesiophobia; Catastrophizing; Anxiety; Depression
MeSH Terms: conditions — Hemophilia A; Arthralgia; Kinesiophobia; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational group: Patients who meet all inclusion criteria will be informed verbally and in writing of the characteristics, objectives, and risks of the intervention. They will be provided with patient information and informed consent documents. After confirming that they do not meet any of the exclusion criteria, the dependent and confounding variables of the study will be evaluated. The evaluation will be carried out at the premises of the member associations of the Spanish Hemophilia Federation. All evaluations will be performed by the same physical therapist, following the same evaluation protocol.

SUMMARY:
Introduction: Hemophilic arthropathy is characterized by functional impairments, disabling physical sequelae, and chronic pain. Central pain sensitization describes increased neural excitability characterized by spontaneous or persistent pain, increased pain areas, allodynia, and hyperalgesia.

Objectives: To evaluate central pain sensitization in patients with hemophilia and degenerative knee and ankle arthropathy and to identify the best predictive model of central pain sensitization in these patients.

Methods: Multicenter cross-sectional cohort study. Eighty-six patients with hemophilic knee and ankle arthropathy will be recruited through the Spanish Hemophilia Federation. The primary outcome measure will be central pain sensitization (Central Sensitization Inventory), with age as the dependent variable. The secondary variables will be kinesiophobia (Tampa Scale for Kinesiophobia), catastrophizing (Pain Catastrophizing Scale), and pain anxiety (Pain Anxiety Symptoms Scale-20). The variables estimated as modifiers or confounders will be pain intensity (Visual Analogue Scale), joint status (Hemophilia Joint Health Score), severity and type of hemophilia, development of inhibitors, and sociodemographic variables.

Expected results: To identify the degree of central pain sensitization in patients with hemophilic arthropathy. To identify the best predictive model for central pain sensitization in these patients based on the study variables.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with haemophilia A and B.
* Over 35 years of age.
* With a medical diagnosis of bilateral haemophilic ankle arthropathy.
* With a clinical assessment using the Hemophilia Joint Health Score greater than 4 points.
* On prophylactic treatment with FVIII/FIX coagulation concentrates or monoclonal antibodies.
* Sign the informed consent document.

Exclusion Criteria:

* Patients with neurological or cognitive impairments that prevent them from understanding the questionnaires and physical tests.
* Patients who have had ankle or knee haemarthrosis in the 6 months prior to the start of the study.
* Patients who have taken analgesic or anti-inflammatory drugs in the 10 days prior to the study.
* Patients who are undergoing an intervention (physiotherapy or orthopaedic) at the time of the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with hemophilia and degenerative knee and ankle arthropathy
Sampling Method: Non-Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-10-28 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of central pain sensitivity at baseline. | Baseline
  The Spanish version of the Central Sensitisation Inventory will be used to assess the presence of central sensitisation in patients. The first part of this inventory consists of 25 items that assess possible healthy symptoms. Each item is assessed using a 5-point Likert scale with a numerical hierarchy: Never (0), Rarely (1), Sometimes (2), Often (3) and Always (4). The second part assesses whether the patient has been diagnosed with any of a list of 10 disorders, including the year of diagnosis. The reliability of this inventory is very high (ICC: 0.82-0.97). The assessment of the first part of this tool ranges from 0 to 100 points, where the higher the score, the greater the clinical severity of the patients.

SECONDARY OUTCOMES:
Assessment of fear of movement at baseline | Baseline
  Fear of movement will be assessed using the Spanish version of the Tampa Scale of Kinesiophobia (TSK-11SV). This scale consists of 11 items, each of which can be scored from 1 to 4. This scale shows high reliability (ICC = 0.87). The score range on the scale is 11 to 44 points, with higher scores indicating greater fear of movement.
Assessment of catastrophising at baseline | Baseline
  The catastrophising of the patients in the study will be measured using the validated Spanish version of the Pain Catastrophising Scale. This scale consists of 13 items, each of which can be scored from 0 to 4. This scale has demonstrated high reliability (ICC = 0.84). The scale ranges from 0 to 52 points, with higher scores indicating greater catastrophising.
Assessment of pain anxiety levels at baseline | Baseline
  The Pain Anxiety Symptoms Scale-20 (PASS-20) will be used to assess levels of anxiety related to pain. This scale has 20 items and measures anxiety and fear responses associated with the experience of chronic or recurrent pain. Each item is rated on a 5-point scale, from 0 (never) to 5 (always). It consists of four domains that measure cognitive anxiety responses, escape and avoidance, fearful thoughts, and physiological anxiety responses. This instrument has shown moderate reliability (CCI= 0.71).

OTHER OUTCOMES:
Assessment of joint pain intensity at baseline | Baseline
  The visual analogue scale will be used to measure perceived joint pain intensity. The score for perceived pain ranges from 0 to 10 points, where 0 is the minimum (no pain) and 10 is the maximum (maximum pain).
Assessment of joint damage at baseline | Baseline
  Joint damage will be measured using the Haemophilia Joint Health Score (HJHS) tool. This scale is designed to identify joint degeneration in the elbows, knees and ankles in children, adolescents and adults with haemophilia. It consists of eight items: inflammation and its duration, pain, muscle atrophy and strength, crepitus, and loss of flexion and extension. This tool has good reliability (ICC > 70). Scores range from 0 to 20 points (maximum joint damage) per joint. To assess total joint damage, a gait assessment (range 0-4 points) is added, with a maximum score of 124 points.
Assessment of the sociodemographic variable age at baseline | Baseline
  The sociodemographic variable age will be measured in months completed from the patient's date of birth to the date of the assessment.
Assessment of the sociodemographic variable marital status at baseline | Baseline
  The sociodemographic variable marital status will be measured using 4 response options (qualitative variable): single / married / divorced / widowed.
Assessment of the clinical variable type of haemophilia at baseline | Baseline
  The clinical variable type of haemophilia will be measured using a dichotomous qualitative variable with two response options: haemophilia A / haemophilia B.
Assessment of the clinical variable severity of haemophilia at baseline | Baseline
  The clinical variable severity of haemophilia will be measured using a qualitative variable with three response options: mild/moderate/severe.
Assessment of the clinical variable development of inhibitors at baseline | Baseline
  The clinical variable development of inhibitors to clotting factor concentrates will be measured using a dichotomous qualitative variable with two response options: yes/no.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Universidad de Oviedo
Locations (1):
- Universidad de Oviedo, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: No